CLINICAL TRIAL: NCT01807520
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Study to Demonstrate the Efficacy at 16 Weeks of Secukinumab 150 and 300 mg s.c. and to Assess Safety, Tolerability and Long-term Efficacy up to 132 Weeks in Subjects With Moderate to Severe Nail Psoriasis
Brief Title: Study of Safety, Tolerability, and Efficacy of Secukinumab in Subjects With Moderate to Severe Nail Psoriasis
Acronym: TRANSFIGURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457A2313; 2012-005413-40 (EudraCT Number)
Record Dates: First submitted 2013-01-23; First posted 2013-03-08 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Moderate to Severe Nail Psoriasis
Keywords: Moderate nail psoriasis; Severe nail psoriasis; psoriasis; Secukinumab
MeSH Terms: conditions — Psoriasis | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Secukinumab (AIN457) 150 mg (Experimental): Participants assigned to secukinumab 150 mg were dosed weekly for five weeks, then once every four weeks up to and including Week 132. To maintain the blinding, patients received additional placebo injections at Weeks 17, 18 and 19. All doses of study treatment are administered by sub-cutaneous injections.
  Interventions: Biological: Secukinumab
- Secukinumab (AIN457) 300 mg (Experimental): Participants assigned to secukinumab 300 mg were dosed weekly for five weeks, then once every four weeks up to and including Week 132. To maintain the blinding, patients received additional placebo injections at Weeks 17, 18 and 19. All doses of study treatment are administered by sub-cutaneous injections.
  Interventions: Biological: Secukinumab
- Placebo (Placebo Comparator): Patients assigned to placebo were dosed weekly for five weeks, then at Week 8 and Week 12. At Week 16, placebo patients were randomized in a 1:1 ratio, to receive secukinumab either 150 mg or 300 mg and were dosed weekly for five weeks starting at Week 16, then once every four weeks up to and including Week 132. All doses of study treatment are administered by sub-cutaneous injections.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Secukinumab — Study treatment was provided in pre-filled 1 mL syringes.
  Other Names: AIN457
  Arms: Secukinumab (AIN457) 150 mg; Secukinumab (AIN457) 300 mg
Biological: Placebo — Placebo was provided in pre-filled 1 mL syringes.
  Other Names: placebo secukinumab
  Arms: Placebo

SUMMARY:
This purpose of this study was to demonstrate the efficacy of secukinumab versus placebo on nail psoriasis and to assess long-term efficacy, safety and tolerability of secukinumab.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic moderate to severe plaque type psoriasis for at least 6 months prior to randomization, including significant nail involvement, defined as Nail Psoriasis Severity Index (NAPSI) score ≥16 AND number of fingernails involved ≥4 AND Psoriasis Area and Severity Index (PASI) score ≥12 AND Body Surface Area (BSA) score ≥10%
* Candidates for systemic therapy, i.e. psoriasis inadequately controlled by topical treatment (including super potent topical corticosteroids) and/or phototherapy and/or previous systemic therapy

Exclusion Criteria:

* Forms of psoriasis other than chronic plaque type psoriasis (e.g., pustular psoriasis, palmoplantar pustulosis, acrodermatitis of Hallopeau, erythrodermic and guttate psoriasis)
* Drug-induced psoriasis (e.g. new onset or current exacerbation from β-blockers, calcium channel inhibitors or lithium)
* Ongoing inflammatory skin diseases other than psoriasis or any other disease affecting the fingernails which may potentially confound the evaluation of study treatment effects
* Ongoing use of prohibited treatments (e.g. topical or systemic corticosteroids (CS), UV therapy). Washout periods do apply
* Prior exposure to secukinumab (AIN457) or any other biological drug directly targeting IL-17 or the IL-17 receptor
* Exposure to any investigational drugs within 4 weeks prior to study treatment initiation or within a period of 5 half-lives of the investigational treatment, whichever is longer
* History of hypersensitivity to constituents of the study treatment
* Other protocol-defined inclusion/exclusion criteria do apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2013-06-20 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (37):
- United States (9):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Skokie, Illinois
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, High Point, North Carolina
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Houston, Texas
- Australia (3):
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, East Melbourne, Victoria
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Liège
- Czechia (2):
  - Novartis Investigative Site, Ústí nad Labem, Czech Republic
  - Novartis Investigative Site, Prague
- Denmark (3):
  - Novartis Investigative Site, Arhus C
  - Novartis Investigative Site, Copenhagen NV
  - Novartis Investigative Site, Hellerup
- Germany (5):
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Münster
- Greece (2):
  - Novartis Investigative Site, Heraklion, Crete, GR
  - Novartis Investigative Site, Athens
- Spain (5):
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barakaldo, Vizcaya
  - Novartis Investigative Site, Madrid
- United Kingdom (6):
  - Novartis Investigative Site, London, England
  - Novartis Investigative Site, Staffordshire, Staffordshire
  - Novartis Investigative Site, Dudley, West Midlands
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was made up of 4 periods: screening, treatment period 1, treatment period 2 and post-treatment follow-up.
Pre-assignment Details: In treatment period 1, participants were randomized in a 1:1:1 ratio to secukinumab 150mg, secukinumab 300mg or placebo. In treatment period 2, placebo participants were re-randomized in a 1:1 ratio to secukinumab 150mg or secukinumab 300mg. The follow-up period occurred 8 weeks post treatment period 2 (12 weeks post the last dose of secukinumab).
Groups:
- AIN457 150 mg: Participants assigned to secukinumab 150 mg were dosed weekly for five weeks, then once every four weeks up to and including Week 132. To maintain the blinding, participants received additional placebo injections at Weeks 17, 18 and 19. All doses of study treatment were administered by sub-cutaneous injections.
- AIN457 300 mg: Participants assigned to secukinumab 300 mg were dosed weekly for five weeks, then once every four weeks up to and including Week 132. To maintain the blinding, participants received additional placebo injections at Weeks 17, 18 and 19. All doses of study treatment were administered by sub-cutaneous injections.
- Placebo: Participants who received placebo during treatment period 1
- Placebo - AIN457 150 mg: Participants received placebo weekly for five weeks, and then at Week 8 and Week 12. At Week 16, participants were randomized to receive secukinumab 150 mg and were dosed weekly for five weeks starting at Week 16, and then once every four weeks up to and including Week 132. All doses of study treatment were administered by sub-cutaneous injections.
- Placebo - AIN457 300 mg: Participants received placebo weekly for five weeks, and then at Week 8 and Week 12. At Week 16, participants were randomized to receive secukinumab 300 mg and were dosed weekly for five weeks starting at Week 16, and then once every four weeks up to and including Week 132. All doses of study treatment were administered by sub-cutaneous injections.
- Any AIN457 150 mg: Participants who received AIN457 150 mg during treatment period 1 and/or treatment period 2
- Any AIN457 300 mg: Participants who received AIN457 300 mg during treatment period 1 and/or treatment period 2
Period: Treatment Period 1 (0-16 Weeks)
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg | Any AIN457 150 mg | Any AIN457 300 mg
Started | 67 | 66 | 65 | 0 | 0 | 0 | 0
Full Analysis Set | 67 | 66 | 65 | 0 | 0 | 0 | 0
Safety Set | 67 | 65 | 65 | 0 | 0 | 0 | 0
Completed | 63 | 65 | 58 | 0 | 0 | 0 | 0
Not Completed | 4 | 1 | 7 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 0 | 0 | 0 | 0
Not completed — Protocol deviation | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (16-132 Weeks)
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg | Any AIN457 150 mg | Any AIN457 300 mg
Started | 63 | 65 | 0 | 29 | 29 | 0 | 0
Safety Set | 63 | 65 | 0 | 29 | 29 | 0 | 0
Full Analysis Set | 67 | 66 | 0 | 29 | 29 | 0 | 0
Completed | 38 | 47 | 0 | 22 | 24 | 0 | 0
Not Completed | 25 | 18 | 0 | 7 | 5 | 0 | 0
Not completed — Study terminated | 7 | 4 | 0 | 0 | 2 | 0 | 0
Not completed — Protocol deviation | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-compliant with study treatment | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 5 | 3 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 3 | 3 | 0 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 6 | 0 | 2 | 2 | 0 | 0
Period: Follow-up Period (132-140 Weeks)
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg | Any AIN457 150 mg | Any AIN457 300 mg
Started | 0 | 0 | 2 (These participants discontinued from Treatment Period 1.) | 0 | 0 | 81 (These participants received AIN457150mg during treatment period 1 and/or treatment period 2.) | 76 (These participants received AIN457 300mg during treatment period 1 and/or treatment period 2.)
Completed | 0 | 0 | 2 | 0 | 0 | 77 | 75
Not Completed | 0 | 0 | 0 | 0 | 0 | 4 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Study terminated | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | Total
Number analyzed (Participants) | 67 | 66 | 65 | 198
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.5 (10.94) | 45.1 (12.9) | 43.6 (11.2) | 44.1 (11.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 13 | 38
  Male | 55 | 53 | 52 | 160

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Nail Psoriasis Severity Index (NAPSI) After 16 Weeks of Treatment
Description: The NAPSI is a tool to assess psoriatic nail involvement in patients with nail psoriasis. Each nail is divided with imaginary horizontal and longitudinal lines into quadrants. Each nail is given a score for nail matrix psoriasis (0-4) and nail bed psoriasis (0-4) depending on the presence of any of the features of nail psoriasis in that quadrant. Each nail gets a nail matrix score and a nail bed score, the total of which is the NAPSI score for that nail ranging from 0 to 8. All 10 fingernails are assessed giving a total NAPSI score ranging from 0 to 80. A negative change from baseline indicates improvement. The adjusted mean is presented.
Time Frame: Baseline, 16 weeks
Population: Only participants from the full analysis set (FAS) who had values at both baseline and week 16, were analyzed. The FAS consisted of all randomized participants to whom treatment was assigned. The analysis was based on Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Error); unit: percent change
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 63 | 64 | 56
percent change | -38.4 (4.54) | -46.1 (3.43) | -11.7 (4.28)
Statistical Analysis 1: Comparison: AIN457 150 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed model reapeated measures; Mean Difference (Net) = -26.7, 95% CI 2-sided [-39.1 to -14.3], Standard Error of Mean 6.26
Statistical Analysis 2: Comparison: AIN457 300 mg vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed model repeated measures; Mean Difference (Net) = -34.4, 95% CI 2-sided [-45.2 to -23.5], Standard Error of Mean 5.47

2. Secondary Outcome: Percent Change From Baseline in NAPSI Score
Description: The NAPSI is a tool to assess psoriatic nail involvement in patients with nail psoriasis. Each nail is divided with imaginary horizontal and longitudinal lines into quadrants. Each nail is given a score for nail matrix psoriasis (0-4) and nail bed psoriasis (0-4) depending on the presence of any of the features of nail psoriasis in that quadrant. Each nail gets a nail matrix score and a nail bed score, the total of which is the NAPSI score for that nail ranging from 0 to 8. All 10 fingernails are assessed giving a total NAPSI score ranging from 0 to 80. A negative change from baseline indicates improvement.
Time Frame: baseline, 16 weeks, 132 weeks
Population: Only participants from the full analysis set (FAS) who had values at both baseline and the post-baseline time point, were analyzed. The FAS consisted of all randomized participants to whom treatment was assigned. The analysis was based on Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 67 | 65 | 29 | 29
percent change
  Week 16 | -37.9 (37.32) | -45.3 (27.22) | -15.4 (32.79) | -7.8 (31.77)
  Week 132: number analyzed (Participants) | 67 | 65 | 28 | 29
  Week 132 | -52.9 (42.90) | -70.5 (29.2) | -62.9 (29.05) | -72.7 (22.84)

3. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index 75 (PASI75) and Investigator Global Assessment (IGA Mod 2011) Response 0 or 1 Over Time up to Week 16 of the Treatment Compared to Placebo and Over Time up to Week 132
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4). The IGA scale referred exclusively to the participant's disease at the time of the assessment. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe and 5 = very severe. To be considered IGA responder at any point in time, the patient must have an IGA score of 0 or 1 and have achieved a reduction of at least two points on the IGA scale from baseline.
Time Frame: 16 weeks, 132 weeks
Population: Participants from the FAS, who had evaluable data at a given time point, were analyzed for that time point. The FAS consisted of all randomized participants to whom treatment was assigned. Multiple imputation was applied where the number of evaluable participants was based on a rounded mean number of responders for 500 imputations.
Measure: Number; unit: Percentage of participants
Arm/Group | AIN457 150 mg | AIN457 300 mg
Number analyzed (Participants) | 67 | 65
Percentage of participants
  Week 16, PASI 75 | 76.6 | 87.1
  Week 16, IGA 0/1 | 67.8 | 74.0
  Week 132, PASI 75 | 61.6 | 82.7
  Week 132, IGA 0/1 | 52.2 | 61.2

4. Secondary Outcome: Number of Participants Who Develop Immunogenicity Against Secukinumab
Description: The number of participants who tested positive for anti-secukinumab antibodies. It refers to the number of participants who had no positive values at baseline but developed them only after start of secukinumab treatment. None of the participants had a loss of efficacy and the test was only transiently positive.
Time Frame: Week 132
Population: Participants from the safety set was analyzed. The safety set included all participants who took at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo - AIN457 150 mg | Placebo - AIN457 300 mg
Number analyzed (Participants) | 67 | 65 | 29 | 29
Participants | 2 | 5 | 4 | 3

ADVERSE EVENTS:
Time Frame: up to week 140
Groups:
- Any AIN457 Dose: Participants who received AIN457 150 mg or AIN457 300 mg
Arm/Group | Any AIN457 150 mg | Any AIN457 300 mg | Placebo | Any AIN457 Dose
Serious Adverse Events (participants affected / at risk) | 10/96 | 9/94 | 1/65 | 19/190
Other Adverse Events (participants affected / at risk) | 76/96 | 79/94 | 37/65 | 155/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=96) | Any AIN457 300 mg (N=94) | Placebo (N=65) | Any AIN457 Dose (N=190)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Cataract subcapsular (Eye disorders) | 0 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Eczema impetiginous (Infections and infestations) | 1 | 0 | 0 | 1
Eczema infected (Infections and infestations) | 1 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 1 | 0 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=96) | Any AIN457 300 mg (N=94) | Placebo (N=65) | Any AIN457 Dose (N=190)
Palpitations (Cardiac disorders) | 1 | 3 | 0 | 4
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 0 | 3
Hypothyroidism (Endocrine disorders) | 2 | 1 | 0 | 3
Dry eye (Eye disorders) | 2 | 0 | 0 | 2
Eye irritation (Eye disorders) | 2 | 0 | 0 | 2
Eye pruritus (Eye disorders) | 0 | 2 | 0 | 2
Visual impairment (Eye disorders) | 0 | 2 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 5 | 10
Dyspepsia (Gastrointestinal disorders) | 3 | 5 | 0 | 8
Haemorrhoids (Gastrointestinal disorders) | 2 | 1 | 0 | 3
Loose tooth (Gastrointestinal disorders) | 2 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 3 | 1 | 7
Toothache (Gastrointestinal disorders) | 3 | 1 | 0 | 4
Vomiting (Gastrointestinal disorders) | 3 | 1 | 0 | 4
Fatigue (General disorders) | 4 | 5 | 0 | 9
Influenza like illness (General disorders) | 3 | 1 | 0 | 4
Injection site erythema (General disorders) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 3 | 1 | 1 | 4
Hepatic steatosis (Hepatobiliary disorders) | 2 | 2 | 0 | 4
Seasonal allergy (Immune system disorders) | 2 | 1 | 0 | 3
Bronchitis (Infections and infestations) | 4 | 7 | 0 | 11
Cellulitis (Infections and infestations) | 1 | 3 | 0 | 4
Conjunctivitis (Infections and infestations) | 3 | 4 | 0 | 7
Ear infection (Infections and infestations) | 2 | 1 | 0 | 3
Erysipelas (Infections and infestations) | 2 | 1 | 1 | 3
Fungal skin infection (Infections and infestations) | 2 | 1 | 1 | 3
Gastroenteritis (Infections and infestations) | 6 | 6 | 0 | 12
Herpes zoster (Infections and infestations) | 3 | 3 | 0 | 6
Hordeolum (Infections and infestations) | 2 | 1 | 0 | 3
Influenza (Infections and infestations) | 0 | 6 | 2 | 6
Localised infection (Infections and infestations) | 0 | 3 | 0 | 3
Lower respiratory tract infection (Infections and infestations) | 2 | 3 | 0 | 5
Nasopharyngitis (Infections and infestations) | 25 | 27 | 8 | 52
Onychomycosis (Infections and infestations) | 2 | 1 | 0 | 3
Oral candidiasis (Infections and infestations) | 1 | 3 | 0 | 4
Oral herpes (Infections and infestations) | 2 | 2 | 4 | 4
Otitis externa (Infections and infestations) | 1 | 2 | 0 | 3
Pharyngitis (Infections and infestations) | 2 | 3 | 0 | 5
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 2
Pulpitis dental (Infections and infestations) | 4 | 4 | 1 | 8
Respiratory tract infection (Infections and infestations) | 2 | 2 | 0 | 4
Rhinitis (Infections and infestations) | 2 | 7 | 0 | 9
Sinusitis (Infections and infestations) | 3 | 6 | 0 | 9
Skin infection (Infections and infestations) | 1 | 3 | 0 | 4
Tinea pedis (Infections and infestations) | 5 | 1 | 0 | 6
Tonsillitis (Infections and infestations) | 4 | 4 | 0 | 8
Tooth abscess (Infections and infestations) | 0 | 3 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 15 | 8 | 2 | 23
Urinary tract infection (Infections and infestations) | 3 | 5 | 0 | 8
Viral upper respiratory tract infection (Infections and infestations) | 3 | 2 | 0 | 5
Vulvovaginal candidiasis (Infections and infestations) | 2 | 1 | 0 | 3
Arthropod sting (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 3
Limb injury (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 4
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0 | 3
Weight increased (Investigations) | 0 | 2 | 0 | 2
Gout (Metabolism and nutrition disorders) | 2 | 0 | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 8 | 2 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 7 | 1 | 16
Dactylitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 1 | 2 | 6
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 3
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 3
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 1 | 3
Dizziness (Nervous system disorders) | 3 | 1 | 0 | 4
Headache (Nervous system disorders) | 9 | 10 | 4 | 19
Poor quality sleep (Nervous system disorders) | 2 | 0 | 0 | 2
Sciatica (Nervous system disorders) | 2 | 1 | 0 | 3
Anxiety (Psychiatric disorders) | 6 | 0 | 1 | 6
Depression (Psychiatric disorders) | 3 | 4 | 2 | 7
Insomnia (Psychiatric disorders) | 2 | 3 | 0 | 5
Stress (Psychiatric disorders) | 3 | 0 | 0 | 3
Haematuria (Renal and urinary disorders) | 2 | 1 | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 7 | 2 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 3
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 3
Alopecia areata (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 3
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 4 | 0 | 7
Eczema (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 5
Intertrigo (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3 | 1 | 8
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 16 | 6 | 7 | 22
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 3
Hypertension (Vascular disorders) | 5 | 4 | 0 | 9

LIMITATIONS AND CAVEATS:
The overall study completed. However, in Spain, the study terminated early in accordance with study protocol amendment 1.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.